CLINICAL TRIAL: NCT03507517
Title: Quality Control Project of Secondary Prevention and Treatment of Stroke in Liaoning Province
Brief Title: Quality Control Project of Stroke in Liaoning Province
Status: Completed | Type: Observational
Sponsor: Hui-Sheng Chen (Other)
Responsible Party: Sponsor-Investigator, Hui-Sheng Chen, Professor, General Hospital of Shenyang Military Region
Organization: General Hospital of Shenyang Military Region (Other)
Other Study IDs: 2017275212
Record Dates: First submitted 2017-11-26; First posted 2018-04-25 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Stroke, Ischemic
Keywords: prevention
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To reduce the incidence of stroke and standard the treatment of stroke in Liaoning Province, the present study should be conducted.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke

Exclusion Criteria:

* disagreed patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed with ischemic stroke
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Key Performance Indicator of Secondary Prevention of Stroke in Liaoning Province | 2 years
  The real KPI data such as intravenous thrombolysis number and quality, statin use, anti-platelet drugs, VET prevention, etc

SECONDARY OUTCOMES:
The results of Stroke prevention in Liaoning Province | 2 years
  The real data such as good neurological function outcome, stroke recurrence rate, death rate, etc.

IPD SHARING:
Plan to Share IPD: No